CLINICAL TRIAL: NCT03814408
Title: A Phase I Clinical Trial to Evaluate the Safety of the Infusion of Autologous CD34+ Cells Transduced With a Lentiviral Vector Carrying the FANCA Gene in Pediatric Subjects With Fanconi Anemia Subtype A
Brief Title: A Clinical Trial to Evaluate the Safety of RP-L102 in Pediatric Subjects With Fanconi Anemia Subtype A
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-L102-0418
Record Dates: First submitted 2019-01-14; First posted 2019-01-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Fanconi Anemia Complementation Group A
Keywords: FANCA, FA-A, Fanconi Anemia Subtype A
MeSH Terms: conditions — Fanconi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RP-L102 (Experimental): RP-L102 is a self-inactivating lentiviral vector carrying the therapeutic FANCA gene
  Interventions: Biological: RP-L102

INTERVENTIONS:
Biological: RP-L102 — CD34+ enriched cells from subjects with Fanconi anemia subtype A transduced ex vivo with lentiviral vector carrying the FANCA gene, PGK-FANCA-WPRE

SUMMARY:
The objective of this study is to assess the therapeutic safety and preliminary efficacy of a hematopoietic cell-based gene therapy consisting of autologous CD34+ enriched cells transduced with a lentiviral vector carrying the FANCA gene in subjects with Fanconi anemia subtype A (FA-A).

DETAILED DESCRIPTION:
This is a pediatric open-label Phase 1 clinical trial and will include a safety evaluation and preliminary assessment of the efficacy of hematopoietic gene therapy consisting of autologous CD34+ enriched cells transduced with a lentiviral vector carrying the FANCA gene in subjects with FA-A. CD34+ cells will be transduced ex vivo with the therapeutic lentiviral vector and infused following transduction, without any prior conditioning. After transduction, product quality control evaluations will be carried out in aliquots of the transduced population. Investigational product will be infused via intravenous infusion with no upper or lower limit; a dose of ≥5 x 105 CD34+ cells/kg body weight will be considered optimal.

The active agent is a self-inactivating lentiviral vector carrying the therapeutic FANCA gene and the therapeutic product is subject's autologous HSCs that have been transduced with the lentiviral vector. The vector contains the functional FANCA gene.

ELIGIBILITY:
Inclusion Criteria:

* Fanconi anemia, as diagnosed by chromosomal fragility assay of cultured T-lymphocytes in the presence of DEB or a similar DNA-crosslinking agent.
* Subjects of Fanconi Anemia complementation group A.
* Minimum age: 1 year and a minimum of 8 kg.
* Maximum age: 12 years.
* At least one of the following hematologic parameters below lower limits of normal:

  * Hemoglobin
  * Absolute neutrophils
  * Platelets
* At least 30 CD34+ cells/μL are determined in one BM aspiration within 3 months prior to initiation of CD34+ cell collection.
* If the number of C34+ cells/ μL in BM is in the range of 10-29, PB parameters should meet two of the three following criteria:

  * Hemoglobin: ≥11g/dL
  * Neutrophils: ≥900 cells/μL
  * Platelets: ≥60,000 cells/μL
* Provide informed consent in accordance with current legislation.
* Women of childbearing age must have a negative urine pregnancy test at the baseline visit and accept the use of an effective contraception method during participation in the trial.

Exclusion Criteria:

* Subjects with an available and medically eligible human leukocyte antigen (HLA)-identical sibling donor.
* Evidence of myelodysplastic syndrome or leukemia, or cytogenetic abnormalities predictive of these conditions in BM aspirate analysis. This assessment should be made by valid studies conducted within the 3 months before the subject commences the stem cell mobilization/collection procedures of the clinical trial.
* Subjects with somatic mosaicism associated with stable or improved counts in all PB cell lineages. (If T-lymphocyte chromosomal fragility analysis indicates potential mosaicism, a medically significant decrease in at least one blood lineage over time must be documented to enable eligibility).
* Lansky performance status ≤60%.
* Any concomitant disease or condition that, in the opinion of the Principal Investigator, renders the subject unfit to participate in the study.
* Pre-existing sensory or motor impairment ≥grade 2 according to the NCI CTCAE v5.0 criteria.
* Pregnant or breastfeeding women.
* Hepatic dysfunction as defined by either:

  * Bilirubin >3.0 × upper limit of normal (ULN) or
  * Alanine aminotransferase (ALT) > 5.0 × ULN or
  * Aspartate aminotransferase (AST) > 5.0 × ULN
* Renal dysfunction requiring either hemodialysis or peritoneal dialysis.
* Pulmonary dysfunction as defined by either:

  * Need for supplemental oxygen during the prior 2 weeks in absence of acute infection.
  * Oxygen saturation by pulse oximetry <90%.
* Evidence of active metastatic or locoregionally advanced malignancy for which survival is anticipated to be less than 3 years.
* Subject is receiving androgens (i.e. danazol, oxymethalone).

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v.5.0 | 3 years
  Evaluation of safety associated with treatment with RP-L102

SECONDARY OUTCOMES:
Phenotypic correction of T-lymphocytes in peripheral blood after infusion of RP-L102 | 3 years
  Assessment of the percentage of peripheral blood T-cells with DEB-induced chromosomal aberrations that decreases from over or equal to 50% at 0-2 months post-infusion to less than 50% during months 6-36 post-infusion (confirmed in at least 2 determinations conducted in each interval).
Phenotypic correction of hematopoietic cells in bone marrow after infusion of RP-L102 | 3 years
  During months 6-36 post-infusion, the survival of bone marrow colony forming units to 10nM MMC increases to over or equal to 10% than values determined at 0-2 months post-infusion. (1 determination is considered valid).
Engraftment of gene-corrected hematopoietic cells after infusion of RP-L102 | 3 years
  The level of gene marking of the FANCA-LV provirus in total peripheral blood cells is at least 0.1 vector copy number/nucleated cell during months 6-36 post-infusion. (This should be confirmed in at least 2 determinations conducted at different intervals). An increase in the vector copy number/peripheral blood cell is observed from 0-2 months post-infusion to the 3rd year post-infusion. (This should be confirmed in at least 2 determinations conducted in each interval periods).
Prevention or rescue of bone marrow failure after infusion of RP-L102 | 3 years
  Assessment of the need for treatment of bone marrow failure 6-36 months post-infusion. During the 3rd year post-infusion, peripheral blood parameters: hemoglobin levels, neutrophils, and platelets will be assessed and considered stable if they remain at over or equal to 80% of values determined at pre-treatment evaluation visit or immediately prior to mobilization before the administration of granulocyte-colony stimulating factor.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Czechowicz, MD, Principal Investigator — Stanford University, Stem Cell Transplantation and Regenerative Medicine
Locations (1):
- Stanford University Institute for Stem Cell Biology and Regenerative Medicine Lucille Packard Children's Hospital, Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No